CLINICAL TRIAL: NCT06991374
Title: Combined Burst Mode Versus Torsional Mode Phacoemulsification for Patients With Hard Nuclear Cataract: A Randomized Control Study
Brief Title: Study on the Surgical Strategy of Corneal Endothelial Protection for Hard Nuclear Cataract Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013021; Grant No. 81770907 & No. 82070 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-05-20; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hard Nuclear Cataract; Phacoemulsification Cataract Surgery; Endothelial Cell Density Loss; Central Corneal Thickness
Keywords: Hard nuclear cataract; phacoemulisification mode; ultrasound time; cumulative dissipated energy

STUDY DESIGN:
Intervention Model Description: all individuals scheduled for cataract surgery were randomly allocated to either the combined mode group (Burst Tor+ Burst US, Group A) or the torsional mode group (Linear Tor, Group B), utilizing an online random number generator.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined burst mode (Experimental): combining the torsional and vertical ultrasound under burst mode(Burst Tor+ Burst US) Phacoemulsification mode Brust mode Torsional amplitude 0-90% Longitudinal power 40% Infusion system Gravity fed Bottle height 50-80 cm Vacuum 360 mmHg Aspiration flow rate 30 cm3/min Burst duration 70 ms Off time 50 ms
  Interventions: Procedure: combined burst mode
- torsional mode (Active Comparator): torsional mode under continues mode (Linear Tor) Phacoemulsification mode Continuous mode Torsional amplitude 0-90% Longitudinal power 0 Infusion system Gravity fed Bottle height 50-80 cm Vacuum 360 mmHg Aspiration flow rate 30 cm3/min Burst duration - Off time -
  Interventions: Procedure: torsional mode

INTERVENTIONS:
Procedure: combined burst mode — the combined burst mode is commonly used in cataract phacoemulsification. This study compares whether the two modes have different outcomes in hard nuclear cataract surgery.
  Arms: Combined burst mode
Procedure: torsional mode — the toesional mode is commonly used in cataract phacoemulsification. This study compares whether the two modes have different outcomes in hard nuclear cataract surgery.
  Arms: torsional mode

SUMMARY:
In this study, we compared two types of phacoemulsification commonly used in cataract surgery to evaluate their effect on the prognosis of patients with hard nuclei. This will provide a theoretical basis for selecting a more appropriate cataract surgery modality in practice in hard-nucleus patients.

DETAILED DESCRIPTION:
In this study, we randomized patients into two groups. One group was the combined mode group in burst mode and the other group was the torsional ultrasound group in continuous mode. Cumulative dissipated energy(CDE) and ultrasound time(UST) were recorded during the procedure. Changes in central cornea thickness(CCT) and endothelial cell density(ECD) of the patients were recorded postoperatively during a 3-month follow-up. Intraoperative and postoperative complications were also recorded. The above data were analyzed to compare the effect of both on postoperative corneal recovery in patients with hard nuclei.

ELIGIBILITY:
Inclusion Criteria:

* patients with age-related cataracts that were only classified by Emery-Little as nuclear hardness grade III-V.
* encompassed a minimum dilated pupil diameter of 7 mm or above, as well as a corneal endothelial cell count exceeding 1200/mm^2.
* Corneal morphology is normal and clear
* Informed consent is required prior to enrollment

Exclusion Criteria:

* Those with white cataracts, histories of eye surgery, and eye diseases such as corneal pathology, uveitis, Fuchs' dystrophy, and glaucoma were excluded.
* Exclude those with comorbid ocular and systemic diseases that affect corneal endothelial cell function
* Exclude those with previous intraocular surgery

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density | At 1day, 1week, 1month, 3months postoperatively.
  Endothelial cell density after cataract surgery.
central cornea thickness | At 1day, 1week, 1month, 3months postoperatively.
  central cornea thickness after cataract surgery.
ultrasound time | During cataract surgery
  ultrasound time during phacoemulsification.
cumulative dissipated energy | During cataract surgery
  cumulative dissipated energy during phacoemulsification.

SECONDARY OUTCOMES:
best-corrected distance visual acuity | At 1day, 1week, 1month, 3months postoperatively.
  best-corrected distance visual acuity after cataract surgery
cornea edema | At 1day, 1week, 1month, 3months postoperatively.
  cornea edema after cataract surgery
occlusion | during surgery
  occlusion during phacoemulsification

CONTACTS AND LOCATIONS:
Overall Officials: Yinghong Ji, Phd, Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (1):
- Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan, and Informed Consent Form will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2024.1.26, for 1month
Access Criteria: researchers and public

REFERENCES:
- [Background] Liu Y, Zeng M, Liu X, Luo L, Yuan Z, Xia Y, Zeng Y. Torsional mode versus conventional ultrasound mode phacoemulsification: randomized comparative clinical study. J Cataract Refract Surg. 2007 Feb;33(2):287-92. doi: 10.1016/j.jcrs.2006.10.044. PMID 17276271